CLINICAL TRIAL: NCT04725474
Title: A Phase 1/2, FIH, Two-part, Open-label Clinical Trial of Intravenous (IV) Administration of CTL-002 Given as Monotherapy and/or in Combination With an Anti-PD-1 Checkpoint Inhibitor in Subjects With Advanced-stage, Relapsed/Refractory Solid Tumors (The "GDFATHER"-Trial: GDF-15 Antibody-mediaTed Human Effector Cell Relocation).
Brief Title: First-in-Human Study of the GDF-15 Neutralizing Antibody Visugromab (CTL-002) in Patients With Advanced Cancer (GDFATHER)
Acronym: GDFATHER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTL-002-001
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
Keywords: CTL-002; GDF-15; visugromab

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to a dose level of CTL-002 (Part A) or an expansion cohort (Part B) at the time of their enrollment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Part A; dose escalation): CTL-002 Monotherapy + Checkpoint Inhibitor Combination (Experimental): Up to 5 dose levels with visugromab (CTL-002) administered as IV monotherapy and in combination with a CPI
  Interventions: Biological: visugromab (CTL-002)
- Phase 2 (Part B; expansion): visugromab (CTL-002) + Checkpoint Inhibitor Combination (Experimental): At defined dose level(s) with visugromab (CTL-002)
  Interventions: Biological: visugromab (CTL-002)

INTERVENTIONS:
Biological: visugromab (CTL-002) — monoclonal antibody

SUMMARY:
The Phase 1 part (Part A) is a dose escalation study of IV visugromab (CTL-002, a monoclonal antibody neutralizing GDF-15) as monotherapy and in combination with an approved checkpoint inhibitor (CPI) in patients with advanced solid tumors.

Enrolment into the Ph 1 part is completed.

The Phase 2 parts (Part B) are cohort expansions with visugromab (CTL-002) in combination with a defined CPI at a fixed dose into seven different solid tumor indications.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent, and able to comply with the study procedures and any locally required authorization.
* Male or female aged ≥ 18 years.
* Relapsed/refractory patients with histologically or cytologically confirmed diagnosis of advanced-stage or recurrent cancer (Germany-specific: and have exhausted all standard of care treatments or are not eligible for such treatments)
* Progressed on/relapsed after at least one prior anti-PD-1/PD-L1 treatment
* Biopsy-accessible tumor lesions and willing to undergo triple sequential tumor biopsy (Part A) and dual biopsy (Part B, only for selected cohorts).
* At least 1 radiologically measurable lesion per RECIST V1.1/imRECIST (Part B).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy > 3 months as assessed by the Investigator.
* Adequate organ function (bone marrow, hepatic, renal function and coagulation).

Main Exclusion Criteria:

* Pregnant or breastfeeding.
* Any tumor-directed therapy within 21 days before study treatment.
* Treatment with investigational agent within 21 days before study treatment.
* Radiotherapy within 14 days before study treatment.
* Pre-existing arrhythmia, uncontrolled angina pectoris, uncontrolled heart failure (NYHA) Grade IV, any myocardial infarction/coronary event, CNS-ischemic event and any thromboembolic event at any time < 6 months prior to Screening or presence of any uncontrolled heart failure NYHA Grade III or higher.
* Left ventricular ejection fraction (LVEF) < 50% measured by echocardiogram or MUGA.
* QTcF > 450 ms for men or > 470 ms for women.
* Any active autoimmune requiring systemic immunosuppressive treatments. .
* Any history of non-infectious pneumonitis < 6 months prior to Screening.
* Any active inflammatory bowel disease such as Crohn's disease or ulcerative colitis which are generally excluded or active autoimmunthyroiditis present < 6 months prior to Screening.
* History of CNS disease such as stroke, seizure, encephalitis, or multiple sclerosis (< 6 months prior to Screening).
* Evidence for active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), tuberculosis (TB), or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Parts A & B) | min. 2 months
  Incidence of treatment emergent adverse events in monotherapy and/or combination therapy
Determination of DLT and MTD (Part A) | 28 days
  Assessment of toxicities in monotherapy and/or combination therapy per dose level
Evaluation of clinical efficacy according RECIST (Part B) | min. 6 weeks
  RECIST is measured every 6-8 weeks treatment

SECONDARY OUTCOMES:
Cmax following the first dose of CTL-002 (Part A & B) | 1 day
  PK parameter from serum CTL-002 levels
AUC following the first dose of CTL-002 (Part A & B) | 14 days
  PK parameter from serum CTL-002 levels
Half-life of CTL-002 (Part A & B) | min. 6 weeks
  PK parameter from serum CTL-002 levels
Evaluation of treatment-emergent cytokine/chemokine concentrations (Part A & B) | min. 6 weeks
  Measurement of concentration in peripheral blood
Evaluation of clinical efficacy according RECIST (Part A) | min. 6 weeks
  RECIST is measured every 6-8 weeks during treatment
Evaluation of appetite (Part A) | min. 6 weeks
  Assessment of appetite via quality of life questionnaire
Assessment of Body-Mass-Index (BMI) (kg/m2) (Part A) | min. 6 weeks
  Calculation of BMI in kg/m2 by combining measurement of body weight in kg and body height in cm
Assessment of lumbar vertebra skeletal muscle index (L3SMI) (cm2/m2) (Parts A & B) | min. 6 weeks
  Combining measurement of L3 vertebra skeletal muscle mass via computed tomography (CT) in cm2 and patient height (squared) in m2

CONTACTS AND LOCATIONS:
Overall Officials: Sujata Rao, MD, Study Director — CatylYm GmbH
Locations (13):
- Germany (3):
  - Universitätsklinikum Essen, Westdeutsches Tumorzentrum, Innere Klinik und Poliklinik, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik I, Frankfurt am Main
  - Universitätsklinikum Würzburg, Comprehensive Cancer Center, Würzburg
- Spain (7):
  - Next Oncology, Phase I Unit. IOB - Hospital Quironsalud, Barcelona
  - Hospital Universitari Vall d'Hebron, Institute of Oncology, Barcelona
  - ICMDiM, Hospital Clinic, Barcelona
  - ICO Hospitalet, Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid, Hospital Universitario HM Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Unidad Central de Ensayos Clinicos, Pamplona
- Switzerland (3):
  - University Hospital Basel, Department for Medical Oncology, Basel
  - Kantonsspital St. Gallen, Clinic for Medical Oncology & Hematology, Sankt Gallen
  - University Hospital Zurich, Department of Dermatology, Zurich

IPD SHARING:
Plan to Share IPD: No